CLINICAL TRIAL: NCT04410380
Title: Patient Portal Use by Parents of Spanish-Speaking Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-1545
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-03

CONDITIONS: Patient Engagement
MeSH Terms: conditions — Patient Participation | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electronic tablet (Experimental): Spanish-speaking parents receive electronic tablet and teaching about use
  Interventions: Behavioral: Electronic tablet provision with teaching

INTERVENTIONS:
Behavioral: Electronic tablet provision with teaching — Spanish-speaking parents are provided with an electronic tablet and taught how to use it to access health information for their children.

SUMMARY:
The purpose of this study is to determine whether patient portal access is feasible and useful for Spanish-speaking parents.

Participants will be given an electronic tablet and will be taught how to access their child's medical record and other electronic health resources using the tablet.

ELIGIBILITY:
Inclusion Criteria:

* Be parent/legal guardians of children receiving care in UNC's Children's Clinics
* Have Spanish as preferred language of individual identifying as primary caregiver
* Have never activated MyChart (patient portal)
* Have internet service at home OR ability to easily access internet service
* Have at least one child under age 13

Exclusion Criteria:

* Medically unstable at time of recruitment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-02 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Percent of Parents Activating Patient Portal | 6 months
  To determine patient portal use.

SECONDARY OUTCOMES:
Change in Parent Attitudes Toward Health Information Technology | Baseline, 1 month
  Parent attitudes and perceptions will be assessed by survey at enrollment and 1 month after intervention. Scale name: Reasons to use more health information technology. Range 3-12. Directionality: Higher scores indicate more favorable attitudes toward health information technology

CONTACTS AND LOCATIONS:
Overall Officials: Kori Flower, MD, MS, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No